CLINICAL TRIAL: NCT05296499
Title: Exercise Physiology After Thrombosis (EXERT): a Prospective Single Centre Cohort Study of Cardiovascular and Exercise Physiology in Patients With Previous Venous Thrombosis in the Inferior Vena Cava and Iliofemoral Veins.
Brief Title: EXERT: Exercise Physiology After Thrombosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 254956
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Venous Thrombosis Deep (Limbs); Post Thrombotic Syndrome
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome | interventions — Exercise Test; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Venous outflow obstruction extending to inferior vena cava, symptomatic with dyspnoea: Baseline assessments Post-operative assessments if applicable
  Interventions: Diagnostic Test: Cardiopulmonary exercise test (CPET); Diagnostic Test: Exercise cardiac MRI; Other: 6 minute walk test; Diagnostic Test: Blood tests; Other: Quality of life questionnaires; Other: Repeat baseline assessments; Diagnostic Test: MR venogram
- Venous outflow obstruction extending to inferior vena cava, not symptomatic with dyspnoea: Baseline assessments Post-operative assessments if applicable
  Interventions: Diagnostic Test: Cardiopulmonary exercise test (CPET); Diagnostic Test: Exercise cardiac MRI; Other: 6 minute walk test; Diagnostic Test: Blood tests; Other: Quality of life questionnaires; Other: Repeat baseline assessments; Diagnostic Test: MR venogram
- Unilateral iliac venous outflow obstruction: Baseline assessments Post-operative assessments if applicable
  Interventions: Diagnostic Test: Cardiopulmonary exercise test (CPET); Diagnostic Test: Exercise cardiac MRI; Other: 6 minute walk test; Diagnostic Test: Blood tests; Other: Quality of life questionnaires; Other: Repeat baseline assessments; Diagnostic Test: MR venogram
- Age and sex matched controls: Baseline assessments
  Interventions: Diagnostic Test: Cardiopulmonary exercise test (CPET); Diagnostic Test: Exercise cardiac MRI; Other: 6 minute walk test; Other: Quality of life questionnaires; Other: Repeat baseline assessments

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test (CPET) — Cardiopulmonary exercise testing using cycle ergonomenter
Diagnostic Test: Exercise cardiac MRI — Exercise cardiac MRI using supine cycle, participants exercised to peak workload as determined by CPET
Other: 6 minute walk test — 6MWT
Diagnostic Test: Blood tests — FBC, U&E, LFTS
  Groups: Unilateral iliac venous outflow obstruction; Venous outflow obstruction extending to inferior vena cava, not symptomatic with dyspnoea; Venous outflow obstruction extending to inferior vena cava, symptomatic with dyspnoea
Other: Quality of life questionnaires — SF36, EQ5D, VEINES-QoL/Sym
Other: Repeat baseline assessments — repeat baseline
Diagnostic Test: MR venogram — MRI scan of venous system
  Groups: Unilateral iliac venous outflow obstruction; Venous outflow obstruction extending to inferior vena cava, not symptomatic with dyspnoea; Venous outflow obstruction extending to inferior vena cava, symptomatic with dyspnoea

SUMMARY:
Deep vein thrombosis (DVT) can cause long-term scarring and narrowing of veins. When there is extensive damage to the veins in the legs, groin or abdomen it can affect the way that blood is able to flow back up to the heart. Some patients are left with severe symptoms such as pain, leg swelling and ulcers, and have surgical treatment with nitinol stents to re-open the veins and relieve symptoms. The primary aim of this study is to investigate venous blood flow to the heart during exercise in patients with extensive damage to the veins in the groin and abdomen after DVT, and changes that happen after stenting.

DETAILED DESCRIPTION:
Participants will have cardiopulmonary exercise testing, 6 minute walk test and basic blood tests to establish exercise tolerance and rule out other heart and lung conditions. Exercise cardiac MRI will be used to evaluate cardiac function during exercise. All participants will complete generic and disease specific quality of life questionnaires.

Participants who are having a stenting procedure will repeat assessments 6-8 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

All groups:

->16 years of age

- Consent to participate in the research study and be willing to commit to study requirements, including completion of questionnaires and follow up visits.

Group 1:

* Venous thrombosis/obstruction involving the inferior vena cava >12 months ago.
* Symptoms of exertional dyspnoea reported by patient.
* Judged by the chief investigator as suitable for surgical intervention before recruitment to the study.
* Agree to adhere to therapeutic anticoagulation after surgical intervention.

Group 2:

* Venous thrombosis/obstruction involving the inferior vena cava >12 months ago.
* Under the clinical care of the deep venous service for surveillance of symptoms.

Group 3:

* Unilateral Iliofemoral venous thrombosis /obstruction >12 months ago.
* Judged by the chief investigator as suitable for surgical intervention before recruitment to the study.
* Agree to adhere to therapeutic anticoagulation after surgical intervention.

Exclusion Criteria:

All groups:

* DVT or PE in last 12 months
* Significant or untreated left sided heart disease (eg coronary artery disease, LV dysfunction, valvular abnormalities, congenital heart disease, chronic or paroxysmal arrhythmias)
* Significant or untreated chronic lung disease (eg asthma, COPD, ILD)
* Moderate to severe renal disease
* Moderate to severe liver disease
* Peripheral arterial disease
* Significant neurological or musculoskeletal disease
* Cognitive impairment or learning disabilities
* Pregnant or planning to become pregnant in next 12 months
* Active cancer (primary, metastatic or treated within last 6 months)
* Life expectancy < 2 years or chronic non-ambulatory status.
* Any other contraindication to exercise.
* Any contraindications to MRI scanning
* Inability to provide informed consent or comply with study assessments (e.g. due to cognitive impairment, physical limitations or geographic distance).

Group 4:

All of the above, plus:

* Previous DVT or PE
* Known, or clinical signs of chronic venous disease as judged by the chief investigator e.g. varicose veins, leg ulcers.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with previous deep vein thrombosis /chronic outflow obstruction in the iliofemoral veins and inferior vena cava.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
VO2 max after stenting | 6-8 weeks post surgery
  As determined by cardiopulmonary exercise testing
Peak cardiac output during exercise | 6-8 weeks post surgery
  as determined by exercise cardiac MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided